CLINICAL TRIAL: NCT05217732
Title: Randomized, Double-blind and Placebo-controled Study to Assess the Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of ZX-7101A and Its Food Effect in China Healthy Adult Volunteers
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetics of ZX-7101A and the Food Effect in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ZX-7101A-201
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2022-01

CONDITIONS: Safety Issues; Tolerance; Pharmacokinetics; Food Effect

STUDY DESIGN:
Intervention Model Description: single ascending doses in part 1 and fasting/nonfasting crossover in part 2
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind, placebo-controled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Single dose of ZX-7101A treatment A (Experimental): Administrated as a single oral dose in healthy subjects
  Interventions: Drug: ZX-7101A; Drug: Placebo
- Single dose of ZX-7101A treatment B (Experimental): Administrated as a single oral dose in healthy subjects
  Interventions: Drug: ZX-7101A; Drug: Placebo
- Single dose of ZX-7101A treatment C (Experimental): Administrated as a single oral dose in healthy subjects
  Interventions: Drug: ZX-7101A; Drug: Placebo
- Single dose of ZX-7101A treatment D (Experimental): Administrated as a single oral dose in healthy subjects
  Interventions: Drug: ZX-7101A; Drug: Placebo
- Single dose of ZX-7101A treatment E (Experimental): Administrated as a single oral dose in healthy subjects
  Interventions: Drug: ZX-7101A; Drug: Placebo
- ZX-7101A food effect (Experimental): Administered as a selected, single oral dose of ZX-7101A in fasting state and non-fasting (with food) state.
  Interventions: Drug: ZX-7101A

INTERVENTIONS:
Drug: ZX-7101A — tablet
Drug: Placebo — Tablet
  Arms: Single dose of ZX-7101A treatment A; Single dose of ZX-7101A treatment B; Single dose of ZX-7101A treatment C; Single dose of ZX-7101A treatment D; Single dose of ZX-7101A treatment E

SUMMARY:
Randomized, double-blind and placebo-controled study to assess the safety, tolerability and pharmacokinetics of single ascending doses of ZX-7101A and its food effect in China healthy adult volunteers. The study is composed of 2 parts. Part 1 is to assess the safety, tolerability and pharmacokinetics of a single ascending doses of ZX-7101A tablet. Part 2 is to assess the food effect on ZX-7101A at a selected dose in a cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults age of 18-45 years old
* BMI in the range of 9~26 kg/m2; Bodyweight (male) ≥50kg, Bodyweight (Female) ≥45kg
* In the judgement of the investigator, no clinically relevant abnormalities identified by a detailed medical history and full physical examination including BP and pulse rate measurement, or clinical laboratory tests
* Female subjects of nonchildbearing potential must be not pregnant or lactating. Subjects must consent and comply with the contraception requirement of the study.
* Able to understand the risks involved in the study, and provide written informed consent before the first study-specific procedure
* Able to understand and comply with the study procedures

Exclusion Criteria:

* History of hypersensitivity or allergy to drug or food
* History of clinically significant abnormalities such as metabolic, liver, kidney, blood, lung, cardiovascular, gastrointestinal, urinary, endocrine, neurological, or psychiatric disorders; or in the judgement of the investigator, any medical abnormality that may be a concern to participate the study.
* Tympanic temperature >37.5℃, Pulse >100bmp or <50bmp, Systolic blood pressure ≥140mHg or ≤90mHg, or Diastolic blood pressure ≥90mHg or<50mHg
* Clinically relevant out-of-range baseline of total white cells or absolute neutrophil count
* Total bilirubin >1.5x ULN, AST >1.5 ULN or ALT >1.5ULN
* Estimated glomerular filtration rate (eGFR) <90 mL/min/1.73 m2
* QTc interval > 450ms （ Fridericia's correction ， QTcF=QT/(RR^0.33) ）, QRS>120ms
* Acute respiratory tract infection within 2 weeks
* Any condition possibly affecting drug absorption, e.g. gastrectomy
* Received treatment of any prescription drug or alternative medicine within 4 weeks before first dosing or any nonprescription drug within 2 weeks or 5x half-life, whichever is longer
* Regular alcohol consumption >14units/week I the past 6 months or positive in alcohol breath test
* Use of tobacco or nicotine containing products more than the equivalent of 5 cigarettes per day within 3 months
* Unwilling or unable to restrict the intake of caffeine or alcohol within 72 hours before dosing or during the in-patient observation period
* Use or intake of any known liver enzyme inducer or inhibitor within 14 days
* History of drug abuse or positive urine drug test
* Positive test for Hepatitis C antibody (HCV), Hepatitis B surface antigen (HbsAg), Human immunodeficiency virus (HIV) antibody, or Syphilis antibody at Screening
* Accumulative blood donation >400ml within 3 months or >200ml within 4 weeks or planning to donate during the study
* Pregnancy or lactating at screening
* Having difficulty of drawing blood from vein
* Treatment with an investigational drug or procedure within 3 months
* Received vaccination within 3 months or plan to be received vaccine during the study
* Received any surgical procedure within 3 months at screening
* Any other reason that, in the opinion of the investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse effect (TEAEs) and severe adverse events (SAEs) | Day 1-day15
  safety and tolerability

SECONDARY OUTCOMES:
Peak plama concentration of ZX-7101A | Days 1-15
  To evaluate the maximum observed concentration (Cmax) after single oral dose of ZX-7101A
Area under the plasma concentration of ZX-7101A | Days 1-15
  To evaluate the area under the curve (AUC) plasma-concentration after single oral dose of ZX-7101A
Half-life of ZX-7101A | Days 1-15
  To evaluate the half-life of ZX-7101A after single oral dose of ZX-7101A
Concentration of ZX-7101A in urine | Days 1-15
  To evaluate the concentration at a select treatment after single oral dose of ZX-7101A

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Qin, PhD, Study Director — Zenshine Pharmaceuticals
Locations (1):
- Fudan University affiliated Huashan Hospital, Shanghai, Shanghai Municipality, China